CLINICAL TRIAL: NCT04599192
Title: Prospective Evaluation of Coronary Artery Disease in Women Presenting With Cardiac Ischemia: an Anatomic and Physiologic Study Comparing Fractional Flow Reserve (FFR) and Instantaneous Free-wave Ratio (iFR) on Cardiac Catheterization With Findings of Inducible Ischemia on Non-invasive Stress Imaging
Brief Title: Fractional Flow Reserve and Instantaneous Free-wave Ratio Revascularization Strategies in Women
Acronym: FiRST
Status: Enrolling by invitation | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 2000024865
Record Dates: First submitted 2020-08-12; First posted 2020-10-22 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Coronary Disease; Percutaneous Coronary Intervention; Exercise Test; Myocardial Perfusion Imaging; Cardiac Catheterization
Keywords: WOMEN FiRST; FFR in Women; iFR in Women
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women Presenting with Cardiac Ischemia: Women presenting with cardiac ischemia as indicated by standard of care non-invasive stress testing with cardiac magnetic resonance (CMR), SPECT myocardial perfusion, and PET myocardial perfusion imaging. This cohort of women must also meet the clinical criteria to undergo coronary angiography. Women may be approached for consent either before or after their coronary angiography procedure.
  Interventions: Other: No study intervention

INTERVENTIONS:
Other: No study intervention — The study does not determine any interventions. Any intervention performed during coronary angiography is considered standard of care.

SUMMARY:
A real world study to evaluate outcomes in women based on guideline identified fractional flow reserve (FFR) and instantaneous wave-free ratio (iFR) cutoffs for ischemia (ischemia defined as FFR ≤ 0.80 and iFR ≤ 0.89).

DETAILED DESCRIPTION:
The WOMEN FiRST (FFR iFR Revascularization Strategies Trial) study collects information from enrolled subjects to create a data repository. The data will be used to further elucidate recommendations for PCI of angiographically intermediate lesions (30-90% stenosis) in epicardial lesions in women by comparing FFR and iFR findings to findings of inducible ischemia on existing non-invasive stress imaging studies. Gender comparisons will also be made from archived and published research data sets from studies comprised up to 80% men. Data will also be stored long term for use in future undefined analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Female ≥ 18 years old at signing of informed consent
2. Suspected myocardial ischemia or acute coronary syndrome
3. Indication for non-invasive perfusion imaging study
4. Indication for diagnostic catheterization
5. Eligible for PCI
6. Signed informed clinical procedural consent by subject or by surrogate

Exclusion Criteria:

1. Inability to receive adenosine or regadenoson (for example, severe reactive airway disease, marked hypotension, or advanced atrioventricular block without pacemaker.
2. Severe cardiomyopathy (ejection fraction <30%)
3. Extremely tortuous or calcified coronary arteries precluding FFR/iFR measurements
4. Patients with left main coronary artery disease requiring revascularization
5. Female of child baring age should have negative pregnancy test
6. Subject is pregnant or breast feeding, or planning to become pregnant
7. Contraindication to non-invasive stress imaging including severe claustrophobia, renal disease with GFR <30 where CMR is indication, any metal in the body which is a contraindication to CMR, allergy to gadolinium contrast
8. ICD or PPM

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is not based on self-representation of gender identity
Study Population: Adult female patients (>18 years of age) presenting with suspected myocardial ischemia or acute coronary syndrome for evaluation of ischemia by non-invasive stress testing and coronary angiography.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-04-19 (Actual); Primary Completion 2026-04-10 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Repeat revascularization | 5 years
  Repeat revascularizations will be documented throughout the course of the 5 year follow up period
Non-fatal myocardial infarction | 5 years
  Non-fatal myocardial infarctions will be documented throughout the course of the 5 year follow up period
Non-fatal stroke | 5 years
  Non-fatal strokes will be documented throughout the course of the 5 year follow up period
Cardiovascular death | 5 years
  Cardiovascular related death will be documented throughout the course of the 5 year follow up period

CONTACTS AND LOCATIONS:
Overall Officials: Elissa Altin, MD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine - Section of Cardiology, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gitto, M., Saito Y., Schneider, M., Papoutsidakis, N., Ardito, S., McCarthy, M., Cristea, E., Lansky, A., Altin, E. (2020). Journal of the American College of Cardiology. Discrepancy Between Visually Assessed and Quantitative Coronary Angiography Derived Diameter Stenosis in a Cohort of Women with Stable Coronary Artery Disease, 75(11). https://www.onlinejacc.org/content/75/11_Supplement_1/178
- [Background] Gitto, M., Saito Y., Schneider, M., Papoutsidakis, N., Ardito, S., McCarthy, M., Cristea, E., Lansky, A., Altin, E. (2020). Journal of the American College of Cardiology. Quantitative Flow Ratio According to Three-Dimensional Quantitative Coronary Angiography Defined Severity of Stenosis in a Cohort of Women with Stable Coronary Artery Disease, 75(11). https://www.onlinejacc.org/content/75/11_Supplement_1/177